CLINICAL TRIAL: NCT00209482
Title: A Multi-Center, Randomized, Placebo Controlled, Double Blind Trial of Metformin in Obese Adolescents.
Brief Title: Glaser Obesity Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaser Pediatric Research Network (Network)
Collaborators: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPRN410.PL2.02; NCT00120146 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-10-05 (Estimated); Status verified 2005-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Metformin

INTERVENTIONS:
Drug: glucophage XR

SUMMARY:
This study will determine if the drug metformin, coupled with diet and exercise counseling, will help obese adolescents lose weight.

DETAILED DESCRIPTION:
America is facing an epidemic of obesity among its youth. In the last seven years, there has been a 50% increase in the prevalence of obesity as defined by a Body Mass Index (BMI) > 30 kg/m². For the morbidly obese adult, which is defined as having a BMI > 35 kg/m², mortality is increased by 152 to 279%. In a Veterans Administration study of obese 25-34 year old males, there was a 13-fold excess mortality rate over 7½ years.

As in adults, risks associated with childhood and adolescent obesity include elevated blood pressure and cholesterol levels, predisposing these individuals to cardiovascular disease. In addition, a significant number of obese youth have abnormally high concentrations of insulin, with an attendant increased risk of developing type 2 diabetes mellitus.

Currently, limited options are available to help such individuals. While attempts at lifestyle change (e.g., altering diet and activity level) may have some success in the short term, attempts at maintaining weight loss over the long term often fail. Furthermore, there are no current medications that will safely induce significant weight loss over time.

Metformin is an oral antihyperglycemic, insulin-sensitizing agent that has been used in many countries for treatment of type 2 diabetes for more than 40 years. In March 1995, it was approved by the Food and Drug Administration for the treatment of adult type 2 diabetes. Metformin improves insulin sensitivity and reduces insulin resistance by hepatic and peripheral actions. It does not increase insulin secretion.

Further, metformin decreases hepatic glucose production and results in weight loss. Compared to available drugs that act similarly, only metformin has weight-lowering activity, perhaps by increasing nitric oxide production and improving insulin sensitivity. It is also possible that the mild gastrointestinal side effects of metformin induce weight loss. Metformin is therefore often the agent of choice in obese, type 2 diabetics. In a study of non-diabetic obese adults, treatment with metformin resulted in decreased food intake, and decreased body weight and fat.

This is a randomized, double blind, placebo controlled, multi-center clinical trial. The primary outcome measure that will be used to test the study hypothesis is change in BMI from week 0 to week 52, as well as change in BMI from week 0 to week 100. Approximately 135 potential subjects will be screened at the participating institutions, and an expected 76 subjects will be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 13.00 and 17.99 at week 0 (Baseline).
* Subjects must have a BMI ≥ 95th percentile for age and gender using the CDC data (see Appendix), but must weigh less than 300 pounds (<136 kilograms) when measured during the initial physical exam at week 0 (Baseline). BMI will be calculated as follows; weight in kilograms  [height in meters]2. This cutoff has been established due to the weight-bearing limits of the table used in performing the DXA scan. Once enrolled, if a subject's weight progresses above 300 pounds, s/he may continue in the study whether it is possible to perform DXA or not.
* Completion of informed consent/assent process

Exclusion Criteria:

* Known diabetes as defined by the American Diabetes Association criteria
* Prior drug therapy to treat diabetes or insulin insensitivity, including any form of insulin or insulin analogs; or any oral antidiabetic medication; acarbose, acetohexamide, chlorpropamide, glimepiride, glipizide, glyburide, metformin, pioglitazone, repaglinide, rosiglitazone, tolazamide, tolbutamide or troglitazone.
* Prior use of drugs to aid in weight loss, including but not limited to: Benzphetamine Hcl, Diethylpropion Hcl, Fenfluramine Hcl, Phendimetrazine Tartrate, Phentermine Hcl, Orlistat, Sibutramine Hcl Monohydrate, Didrex, Tenuate, Pondimin, Bontril-SR, Adipex-P, Fastin, Ionamin, Phentrol, Xenical, Meridia.
* Subject is currently taking the following medications at the time of the Screening visit: Cimetidine, amiloride, digoxin, furosemide, morphine, nifedipine, procainamide, ranitidine, triamterene, trimethoprim, vancomycin and quinidine, as these medications may increase metformin levels.
* Subjects will be excluded from the study if they have taken prescription-strength glucocorticoids (by any route) within three months of the screening visit. Topical glucocorticoids are acceptable if their strength is no greater than the equivalent of 1% hydrocortisone cream.
* History of any syndrome or medical disorder associated with significant obesity, including but not limited to: Prader Willi Syndrome, Bardet-Biedl Syndrome, Cohen Syndrome, Cushing syndrome or disease.
* Prior surgical therapy for obesity
* Subject to be excluded if s/he has attended a formal weight loss program within 6 months prior to the Screening visit.
* In the 6 months prior to Screening, subject has consumed alcohol more frequently than twice per week and/or subject has had more than three alcohol-containing beverages in a 24 hour period.
* Elevated creatinine (> 1.2 mg/dl)
* Untreated disorders of thyroid function
* Elevated liver enzymes (Alanine Aminotransferase [ALT] or Aspartate Aminotransferase [AST]) > 80 (approximately 2 times upper limit of normal)
* Mobility impairment that prevents full participation in recommended physical activity
* Other serious medical condition that the Principal Investigator or Lead Site Investigator determines may put the patient at undue risk if enrolled in the study
* Unable to comply with the protocol in the opinion of the Principal Investigator or the Lead Site Investigator
* Subjects with child-bearing potential who are unwilling to remain abstinent or use an effective method of birth control
* Previous pregnancy

Ages: 13 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 76
Dates: Start 2003-10; Study Completion 2007-11

PRIMARY OUTCOMES:
The primary outcome measure that will be used to test the study hypothesis is change in Body Mass Index (BMI). The mean change from baseline in individual BMIs between the two groups will be compared at two time-points; at week 52 and week 100.

CONTACTS AND LOCATIONS:
Overall Officials: Darrell M Wilson, MD, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Children's Hospital, Boston, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Wilson DM, Abrams SH, Aye T, Lee PD, Lenders C, Lustig RH, Osganian SV, Feldman HA; Glaser Pediatric Research Network Obesity Study Group. Metformin extended release treatment of adolescent obesity: a 48-week randomized, double-blind, placebo-controlled trial with 48-week follow-up. Arch Pediatr Adolesc Med. 2010 Feb;164(2):116-23. doi: 10.1001/archpediatrics.2009.264. PMID 20124139
- [Derived] Lenders CM, Feldman HA, Von Scheven E, Merewood A, Sweeney C, Wilson DM, Lee PD, Abrams SH, Gitelman SE, Wertz MS, Klish WJ, Taylor GA, Chen TC, Holick MF; Elizabeth Glaser Pediatric Research Network Obesity Study Group. Relation of body fat indexes to vitamin D status and deficiency among obese adolescents. Am J Clin Nutr. 2009 Sep;90(3):459-67. doi: 10.3945/ajcn.2008.27275. Epub 2009 Jul 29. PMID 19640956